CLINICAL TRIAL: NCT01472302
Title: Effect of a Closed Loop Ventilation Strategy on Reducing the Total Duration of Mechanical Ventilation of Intubated Intensive Care Unit Patients: A Randomized Controlled Trial
Brief Title: Closed Loop Ventilation Strategy in Intensive Care Unit (ICU) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Cenk Kirakli, Principal investigator, Director of ICU, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IGCEAH-ICU 2
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Respiratory Failure; All Intubated Patients
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASV (Experimental): Adaptive Support Ventilation
  Interventions: Device: Adaptive Support Ventilation
- PCV (Active Comparator): Pressure Controlled Ventilation
  Interventions: Device: Pressure Controlled Ventilation

INTERVENTIONS:
Device: Adaptive Support Ventilation — Ventilation protocol according to the patients ideal body weight
  Arms: ASV
Device: Pressure Controlled Ventilation — Ventilation protocol (6-8 ml/kg tidal volume) according to our ICU
  Arms: PCV

SUMMARY:
Adaptive support ventilation (ASV) is a closed loop ventilation mode that can act both like PCV and PSV automatically. Some studies suggest that ASV can reduce the weaning time in ICU patients. The investigators hypothesized that using ASV from the beginning of intubation can reduce the total duration of MV and LOS in the ICU when compared to conventional modes such as PCV+PSV

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated ICU patients for more than 24 hours

Exclusion Criteria:

* Patient with a tracheostomy
* Patients under home mechanical ventilation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Kirakli, MD, Principal Investigator — Izmir Dr. Suat Seren Chest Diseases and Surgery Training Hospital
Locations (1):
- Izmir Chest Diseases and Surgery Education and Research Hospital, Intensive Care Unit, Izmir, Yenisehir, Turkey (Türkiye)

REFERENCES:
- [Derived] Kirakli C, Naz I, Ediboglu O, Tatar D, Budak A, Tellioglu E. A randomized controlled trial comparing the ventilation duration between adaptive support ventilation and pressure assist/control ventilation in medical patients in the ICU. Chest. 2015 Jun;147(6):1503-1509. doi: 10.1378/chest.14-2599. PMID 25742308